CLINICAL TRIAL: NCT01085630
Title: Randomized Phase II Study of Maintenance Pemetrexed Versus Observation for Patients With Malignant Pleural Mesothelioma Without Progression After First-Line Chemotherapy
Brief Title: Pemetrexed Disodium/Observation in Treating Patients W/ Malignant Pleural Mesothelioma w/Out Progressive Disease After 1st Line Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-30901; CALGB-30901; U10CA180821 (NIH); U10CA031946 (NIH); CDR0000667496 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2010-03-11; First posted 2010-03-12 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Malignant Mesothelioma
Keywords: epithelial mesothelioma; sarcomatous mesothelioma; stage II malignant mesothelioma; stage III malignant mesothelioma; stage IV malignant mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant; Solitary Fibrous Tumor, Pleural | interventions — Pemetrexed; Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Experimental): Patients receive pemetrexed disodium IV over 10 minutes on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: pemetrexed disodium
- Arm II (Active Comparator): Patients undergo observation until disease progression.
  Interventions: Other: clinical observation

INTERVENTIONS:
Drug: pemetrexed disodium — Given IV
  Other Names: 150399-23-8
  Arms: Arm I
Other: clinical observation
  Arms: Arm II

SUMMARY:
RATIONALE: Pemetrexed disodium may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This randomized phase II trial is studying how well pemetrexed disodium or observation works in treating patients with malignant pleural mesothelioma without progressive disease after first-line chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine if maintenance therapy with pemetrexed disodium versus observation improves progression-free survival of patients with malignant pleural mesothelioma who have at least stable disease after completion of first-line therapy comprising pemetrexed disodium with cisplatin or carboplatin.

Secondary

* To determine the overall survival of patients treated with this regimen versus observation.
* To evaluate the frequency of responses in patients treated with this regimen.
* To assess the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to first-line chemotherapy regimen (cisplatin/pemetrexed disodium vs carboplatin/pemetrexed disodium), histologic subtype (epithelioid vs other) and number of courses received (< 6 vs 6).

* Arm I: Patients receive pemetrexed disodium IV over 10 minutes on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients undergo observation until disease progression. After completion of study therapy, patients are followed up every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignant pleural mesothelioma meeting 1 of the following cell types:

  * Epithelial
  * Sarcomatoid
  * Mixed type

    * Histologically documented malignant pleural mesothelioma, epithelial, sarcomatoid or mixed type, not amenable to surgical resection
    * Prior treatment
* Currently receiving first-line treatment with pemetrexed + platinum; patients are to be registered to Cancer and Leukemia Group B (CALGB) 30901 no later than the last day of cycle 4 of first line therapy
* Prior intracavitary cytotoxic or sclerosing therapy (including bleomycin) are acceptable; prior intrapleural cytotoxic chemotherapy will not be considered systemic chemotherapy
* Prior surgical treatment is allowed
* Prior radiation therapy is allowed

  * Non-pregnant and non-nursing; women of child bearing potential and men must agree to use an appropriate method of birth control throughout their participation in this study; appropriate methods of birth control include abstinence, oral contraceptives, implantable hormonal contraceptives (Norplant), or double barrier methods (diaphragm plus condom)
  * RANDOMIZATION ELIGIBILITY CRITERIA
  * Patients with complete response, partial response, or stable disease following 4, 5 or 6 cycles of first-line chemotherapy with pemetrexed AND either cisplatin or carboplatin; a maximum of 6 cycles of chemotherapy may have been given
  * Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
  * Granulocytes >= 1,500/ul
  * Platelet count >= 100,000/ul
  * Total bilirubin =< 1.5 x upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) =< 2 x ULN
  * Calculated creatinine clearance >= 45 ml/min
* Disease not amenable to surgery
* Must be enrolled on imaging protocol CALGB-580903
* Complete response, partial response, or stable disease after completion of 4 courses of first-line chemotherapy comprising pemetrexed disodium AND cisplatin or carboplatin

  * Study therapy will begin within 9 weeks following day 1 of cycle 4 of first-line treatment
* No clinically significant pleural or peritoneal effusions that cannot be adequately managed by drainage before or during pemetrexed disodium

PATIENT CHARACTERISTICS:

* ECOG performance status of 0-1
* Life expectancy ≥ 12 weeks
* Granulocytes ≥ 1,500/μL
* Platelet count ≥ 100,000/μL
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST ≤ 2 times ULN
* Creatinine clearance ≥ 45 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No psychiatric illness that would prevent the patient from giving informed consent
* No second malignancy except non-melanoma skin cancer or carcinoma in situ of the cervix unless curatively treated with no evidence of active disease for ≥ 5 years
* No medical conditions that, in the opinion of the treating physician, would make study treatment unreasonably hazardous for the patient including, but not limited to, the following:

  * Ongoing or active infection such as HIV positivity
  * Inability to take oral medications
  * Psychiatric illness/social situations that would limit compliance with study requirements

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior intracavitary cytotoxic or sclerosing therapy (including bleomycin) allowed

  * Prior intrapleural cytotoxic chemotherapy not considered systemic chemotherapy
* Prior surgery allowed
* Prior radiotherapy allowed

  * No concurrent palliative radiotherapy
* No concurrent hormones or other chemotherapeutic agents except for the following:

  * Steroids for adrenal failure
  * Hormones for nondisease-related conditions (e.g., insulin for diabetes)
  * Intermittent use of dexamethasone as an antiemetic or premedication for pemetrexed disodium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2021-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arkadiusz Dudek, MD, Study Chair — Masonic Cancer Center, University of Minnesota
Locations (145):
- United States (145):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - George Bray Cancer Center at the Hospital of Central Connecticut - New Britain Campus, New Britain, Connecticut
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - La Grange Memorial Hospital, La Grange, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - OSF Holy Family Medical Center, Monmouth, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Michiana Hematology-Oncology, PC - Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - Michiana Hematology Oncology PC - Plymouth, Plymouth, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC - La Porte, Westville, Indiana
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - McPherson, McPherson, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Ochsner Health Center - Bluebonnet, Baton Rouge, Louisiana
  - Ochsner Health Center - Covington, Covington, Louisiana
  - New Orleans Cancer Institute at Memorial Medical Center, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Veterans Affairs Medical Center - Baltimore, Baltimore, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - St. Joseph's Medical Center, Brainerd, Minnesota
  - Essentia Health - Duluth Clinic, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Duke Cancer Institute, Durham, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Barberton Citizens Hospital, Barberton, Ohio
  - Cleveland Clinic Beachwood Family Health and Surgery Center, Beachwood, Ohio
  - Cleveland Clinic Cancer Center at Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Cleveland Clinic Cancer Center, Independence, Ohio
  - Hillcrest Cancer Center at Hillcrest Hospital, Mayfield Heights, Ohio
  - Parma Community General Hospital, Parma, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Cleveland Clinic Foundation - Strongsville, Strongsville, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Willamette Falls Hospital, Oregon City, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Roper St. Francis Cancer Center at Roper Hospital, Charleston, South Carolina
  - Danville Regional Medical Center, Danville, Virginia
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Northwest Cancer Specialists at Vancouver Cancer Center, Vancouver, Washington
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 19 enrolled patients were not randomized for the following reasons: progression during first-line therapy, patient refusal, new disease grade 4 brain tumor, patient expired prior to randomization, insufficient creatinine levels, > 1 week needed to randomize, prolonged adverse events, ineligible due to ECOG performance status being 2 or 3.
Groups:
- Arm A (Observation): Patients undergo observation until disease progression.
- Arm B (Pemetrexed): Patients receive pemetrexed 500 mg/m2 IV over 10 minutes (or per institutional guidelines) every three weeks. Patients will continue treatment until disease progression or excess toxicity.
Period: Overall Study
Arm/Group | Arm A (Observation) | Arm B (Pemetrexed)
Started | 26 | 27
Completed | 22 | 27
Not Completed | 4 | 0
Not completed — Insufficient data | 1 | 0
Not completed — Ineligible | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Observation) | Arm B (Pemetrexed) | Total
Number analyzed (Participants) | 22 | 27 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.1 (10.2) | 71.0 (9.0) | 69.7 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 15 | 21 | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Unknown | 1 | 3 | 4
  White | 21 | 23 | 44
  Black/African American | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 27 | 49
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group PS Scale: 0)Fully active, able to carry on all pre-disease performance without restriction; 1)Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2)Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; 3)Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4)Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.
  Participants
    0 | 6 | 9 | 15
    1 | 16 | 18 | 34

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression free survival (PFS) is defined as the time from the date of randomization to the date of disease progression or death resulting from any cause, whichever comes first. Progression is defined according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. The median and 95% confidence intervals are estimated using the Kaplan-Meier estimator.
Time Frame: Baseline up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Observation) | Arm B (Pemetrexed)
Number analyzed (Participants) | 22 | 27
months | 3.0 [2.6 to 11.9] | 3.4 [2.8 to 9.8]

2. Secondary Outcome: Overall Survival
Description: Overall survival time is defined as the time from randomization to death due to any cause. The median and 95% confidence intervals are estimated using the Kaplan-Meier estimator.
Time Frame: Baseline up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Observation) | Arm B (Pemetrexed)
Number analyzed (Participants) | 22 | 27
months | 11.8 [9.3 to 28.7] | 16.3 [10.5 to 26.0]

3. Secondary Outcome: Response Rate
Description: The response rate (percentage) is the percent of patients whose best response was Complete Response (CR) or Partial Response (PR) as defined by RECIST 1.1 criteria. Percentage of successes will be estimated by 100 times the number of successes divided by the total number of evaluable patients. Response rates (including complete and partial response) will be tested using Fisher's exact test
Time Frame: Up to 3 years
Population: One patient on the observation arm did not submit any follow-up forms and withdrew consent to all follow-up and thus excluded in this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (Observation) | Arm B (Pemetrexed)
Number analyzed (Participants) | 21 | 27
percentage of participants | 0 [0 to 0] | 11.1 [2.4 to 29.2]
Statistical Analysis 1: Comparison: Arm A (Observation) vs Arm B (Pemetrexed); Test type: Superiority; p = 0.2423, Fisher Exact

4. Secondary Outcome: Toxicity, Assessed Using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 (v4)
Description: The number of patients reporting grade 3 or higher adverse events considered at least possibly related to study treatment as graded by the NCI's Common Toxicity Criteria (CTCAE) Version 4 are reported here. A complete list of all reported adverse events is reported in the Adverse Events section of this report.
Time Frame: Baseline up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm B (Pemetrexed)
Number analyzed (Participants) | 27
Participants
  Grade 3 Adverse Event | 9
  Grade 4 Adverse Event | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected at the end of each cycle for patients randomized to the treatment arm; Up to 3 years.
Description: Each CTCAE term is a unique representation of a specific event used for medical documentation and scientific analysis and is a single MedDRA Lowest Level Term (LLT). All graded AEs are reported for patients who received treatment (pemetrexed). Serious AE (SAE) reports may include any secondary serious or non-serious events considered related to the primary event (the reason for filing an expedited report); collectively, these events are referred to as Expedited AEs, and appear in the SAE table.
Arm/Group | Arm B (Pemetrexed)
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 3/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm B (Pemetrexed) (N=27)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (2)
Skin infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 2 (2)
INR increased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (2)
Anxiety (Psychiatric disorders) | 1 (2)
Proteinuria (Renal and urinary disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm B (Pemetrexed) (N=27)
Anemia (Blood and lymphatic system disorders) | 18 (101)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (3)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Eyelid function disorder (Eye disorders) | 1 (2)
Watering eyes (Eye disorders) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (10)
Bloating (Gastrointestinal disorders) | 1 (16)
Constipation (Gastrointestinal disorders) | 7 (56)
Diarrhea (Gastrointestinal disorders) | 4 (14)
Dry mouth (Gastrointestinal disorders) | 1 (14)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (4)
Hemorrhoids (Gastrointestinal disorders) | 1 (2)
Mucositis oral (Gastrointestinal disorders) | 3 (13)
Nausea (Gastrointestinal disorders) | 13 (88)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (9)
Chills (General disorders) | 1 (3)
Edema limbs (General disorders) | 4 (13)
Fatigue (General disorders) | 22 (170)
Fever (General disorders) | 2 (3)
Infusion site extravasation (General disorders) | 2 (2)
Localized edema (General disorders) | 2 (10)
Non-cardiac chest pain (General disorders) | 4 (23)
Pain (General disorders) | 6 (10)
Anorectal infection (Infections and infestations) | 1 (6)
Bronchial infection (Infections and infestations) | 1 (1)
Eye infection (Infections and infestations) | 1 (2)
Lung infection (Infections and infestations) | 1 (2)
Prostate infection (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 2 (14)
Tooth infection (Infections and infestations) | 2 (3)
Fall (Injury, poisoning and procedural complications) | 1 (3)
Alanine aminotransferase increased (Investigations) | 5 (14)
Alkaline phosphatase increased (Investigations) | 3 (10)
Aspartate aminotransferase increased (Investigations) | 3 (5)
CD4 lymphocytes decreased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 5 (11)
GGT increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 8 (68)
Lymphocyte count increased (Investigations) | 1 (3)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 3 (6)
Weight gain (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 2 (18)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 5 (8)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (72)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (9)
Hypernatremia (Metabolism and nutrition disorders) | 1 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (37)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (7)
Hyponatremia (Metabolism and nutrition disorders) | 4 (26)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (6)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (8)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (14)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (4)
Dizziness (Nervous system disorders) | 4 (15)
Peripheral motor neuropathy (Nervous system disorders) | 1 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (31)
Anxiety (Psychiatric disorders) | 2 (27)
Insomnia (Psychiatric disorders) | 1 (13)
Chronic kidney disease (Renal and urinary disorders) | 1 (5)
Proteinuria (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (46)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (8)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (14)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (19)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (5)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (5)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (3)
Hot flashes (Vascular disorders) | 1 (21)
Hypertension (Vascular disorders) | 2 (25)
Hypotension (Vascular disorders) | 1 (2)
Thromboembolic event (Vascular disorders) | 2 (5)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-03): https://cdn.clinicaltrials.gov/large-docs/30/NCT01085630/Prot_SAP_000.pdf